CLINICAL TRIAL: NCT01426438
Title: Effect of HDL-Raising Therapies on Endothelial Function, Lipoproteins, and Inflammation in HIV-infected Subjects With Low HDL Cholesterol: A Phase II Randomized Trial of Extended Release Niacin vs. Fenofibrate
Brief Title: Endothelial Function, Lipoproteins, and Inflammation With Low HDL Cholesterol in HIV: ER Niacin Versus Fenofibrate
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5293; 1U01AI068636 (NIH)
Record Dates: First submitted 2011-08-30; First posted 2011-08-31 (Estimated); Results first posted 2014-10-21 (Estimated); Last update posted 2016-02-03 (Estimated); Status verified 2016-01

CONDITIONS: HIV-1 Infection
MeSH Terms: interventions — Niacin; Aspirin; Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Extended-release niacin with aspirin (Experimental)
  Interventions: Drug: Niacin; Drug: Aspirin
- Arm B: Fenofibrate (Experimental)
  Interventions: Drug: Fenofibrate

INTERVENTIONS:
Drug: Niacin — Extended-release niacin will be given with aspirin 325 mg by mouth in the evening and dose-escalated as follows: 500 mg once daily for 4 weeks, 1000 mg once daily for 4 weeks, then 1500 mg once daily for 16 weeks (through week 24)
  Arms: Arm A: Extended-release niacin with aspirin
Drug: Aspirin — Aspirin 325 mg will be given by mouth in the evening with extended-release niacin through week 24.
  Arms: Arm A: Extended-release niacin with aspirin
Drug: Fenofibrate — Fenofibrate will be administered as 200 mg by mouth once daily for 24 weeks.
  Arms: Arm B: Fenofibrate

SUMMARY:
This study is being done with people with HIV infection who have low levels of HDL-C. HDL-C is a type of "good" cholesterol. People with low HDL-C have a higher risk of heart disease and may have problems with how their blood vessels relax. The endothelium is the inner lining of all blood vessels, such as arteries and veins. When the endothelium is not working properly, the blood vessels have trouble expanding properly, which contributes to the development of heart and blood vessel disease.

The main purpose of this study is to see if taking either extended-release niacin or fenofibrate for 24 weeks will help blood vessels work better by improving endothelial function and increasing HDL-C. Niacin and fenofibrate are medications that raise HDL-C. This study will also help determine how safe extended-release niacin and fenofibrate are.

The analysis is an as-treated analysis of participants who completed study treatment and had a week 24 BART scan. Safety analyses include all participants

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* Currently on continuous ART for ≥48 weeks.
* CD4+ cell count ≥100/mm3 obtained within 60 days prior to study entry.
* Most recent HIV-1 RNA below the limit of detection using an ultrasensitive licensed or FDA-approved assay obtained within 60 days prior to study entry.
* Certain laboratory values obtained within 60 days prior to study entry (as indicated in the protocol).
* HDL-C ≤ 40 mg/dL for men or ≤ 50 mg/dL for women within 60 days prior to study entry by any local assay.
* Fasting triglycerides 150-800 mg/dL within 60 days prior to study entry, (initially 200-800 mg/dL, amended during study conduct).
* LDL-C < 160 mg/dL within 60 days prior to study entry.
* For women of reproductive potential, negative serum or urine pregnancy test with a sensitivity of 15-25 mIU/mL within 60 days prior to entry.
* Female subjects of reproductive potential must agree to use a reliable method of contraception while receiving study drug and for 6 weeks after stopping study drug.

Exclusion Criteria:

* Anticipation of changing ART.
* Intent to initiate or change the dose of lipid-lowering drugs or antihypertensives during study.
* Active acute infection or other serious illness requiring systemic treatment and/or hospitalization until subject either completes or is clinically stable on therapy in the opinion of the site investigator.
* Untreated hypogonadism
* History of physician-diagnosed diabetes mellitus or currently taking glucose-lowering medication, (amended during study conduct to allow well-controlled diabetics who are diet controlled or on stable antidiabetic treatment of metformin, sulfonylurea, meglitinides or alpha-glucosidase inhibitors).
* Hormonal anabolic therapies within 90 days prior to study entry.
* Uncontrolled hypertension within 60 days of study entry.
* Acute symptoms of gout within 60 days prior to study entry.
* Active peptic ulcer disease as defined by a health care professional. Treatment for gastroesophageal reflux disease (GERD) is not exclusionary.
* Documented untreated hypothyroidism per subject's medical records.
* Use of thyroid hormone supplements other than for treatment of hypothyroidism within 30 days prior to entry.
* Active or symptomatic gallbladder disease within 1 year of study entry.
* Active cancer requiring systemic chemotherapy or radiation within 1 year of study entry.
* Lipid-lowering agents within 30 days prior to study entry.
* Use of fish oil with DHA/EPA >1000 mg/day within 30 days prior to entry.
* Niacin or niacin-containing products that contain >100 mg daily within 30 days prior to study entry.
* Use of vitamin E supplements greater than 200 IU/day within 30 days prior to entry.
* Use of vitamin C supplements greater than 250 mg/day within 30 days prior to entry.
* Use of systemic cancer chemotherapy, immunomodulators (e.g., growth factors, immune globulin, interleukins, and interferons) within 90 days prior to study entry.
* Any systemic glucocorticoid above replacement levels, defined as the equivalent of ≥ 7.5 mg of prednisone daily, within 60 days prior to study entry.
* Allergy, sensitivity, or severe intolerance to both aspirin and naproxen (Aleve, Naprosyn).
* Symptomatic pancreatitis with hospitalization.
* Pregnancy or currently breastfeeding.
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements.
* Currently taking or anticipation of starting medication during the study for hepatitis C including interferon and ribavirin.
* Documented history of macular edema.
* Current severe congestive heart failure (New York Heart Association [NYHA] Class III or IV).
* History of or current diagnosis of coronary artery disease, angina pectoris, myocardial infarction, previous coronary artery intervention (stenting, angioplasty), peripheral arterial disease (claudication, peripheral arterial angioplasty, or peripheral arterial bypass procedure), cerebrovascular disease (stroke or transient ischemic attack with documented carotid or aortic atherosclerosis), or abdominal aortic aneurysm.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 99 (Actual)
Dates: Start 2011-11; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Dube, MD, Study Chair — University of Southern California; James H Stein, MD, Study Chair — University of Wisconsin School of Medicine and Public Health (Northwestern University CRS)
Locations (14):
- United States (14):
  - Alabama Therapeutics CRS (5801), Birmingham, Alabama
  - University of Southern California (1201), Los Angeles, California
  - UCLA CARE Center CRS (601), Los Angeles, California
  - Harbor-UCLA Med. Ctr. CRS (603), Torrance, California
  - University of Colorado Hospital CRS (6101), Aurora, Colorado
  - Northwestern University CRS (2701), Chicago, Illinois
  - New Jersey Medical School-Adult Clinical Research Ctr. CRS (31477), Newark, New Jersey
  - NY Univ. HIV/AIDS CRS (401), New York, New York
  - Unc Aids Crs (3201), Chapel Hill, North Carolina
  - Duke Univ. Med. Ctr. Adult CRS (1601), Durham, North Carolina
  - Moses H. Cone Memorial Hospital CRS (3203), Greensboro, North Carolina
  - Univ. of Cincinnati CRS (2401), Cincinnati, Ohio
  - Case CRS (2501), Cleveland, Ohio
  - University of Washington AIDS CRS (1401), Seattle, Washington

REFERENCES:
- [Background] International Conference on Harmonisation. E2A: Clinical Safety Data Management : Definitions and Standards for Expedited Reporting. Website: http://www.ich.org/products/guidelines/efficacy/efficacy-single/article/clinical-safety-data-management-definitions-and-standards-for-expedited-reporting.html. Accessed May 24, 2011.
- [Derived] Dube MP, Chan ES, Lake JE, Williams B, Kinslow J, Landay A, Coombs RW, Floris-Moore M, Ribaudo HJ, Yarasheski KE. A Randomized, Double-blinded, Placebo-controlled Trial of Sitagliptin for Reducing Inflammation and Immune Activation in Treated and Suppressed Human Immunodeficiency Virus Infection. Clin Infect Dis. 2019 Sep 13;69(7):1165-1172. doi: 10.1093/cid/ciy1051. PMID 30535188
- [Derived] Dube MP, Komarow L, Fichtenbaum CJ, Cadden JJ, Overton ET, Hodis HN, Currier JS, Stein JH; AIDS Clinical Trials Group A5293 Study Team. Extended-Release Niacin Versus Fenofibrate in HIV-Infected Participants With Low High-Density Lipoprotein Cholesterol: Effects on Endothelial Function, Lipoproteins, and Inflammation. Clin Infect Dis. 2015 Sep 1;61(5):840-9. doi: 10.1093/cid/civ385. Epub 2015 May 15. PMID 25979307

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A5293 opened to accrual under protocol version 1.0 on November 8, 2011. The first participant was enrolled on January 10, 2012. Accrual to the study closed on April 24, 2013, with a total of 99 participants enrolled from 11 sites within the US.
Groups:
- Arm A: Extended-release Niacin With Aspirin: Niacin: Extended-release niacin given with aspirin 325 mg by mouth in the evening and dose-escalated as follows: 500 mg once daily for 4 weeks, 1000 mg once daily for 4 weeks, then 1500 mg once daily for 16 weeks (through week 24)
  Aspirin: Aspirin 325 mg given by mouth in the evening with extended-release niacin through week 24.
- Arm B: Fenofibrate: Fenofibrate: Fenofibrate administered as 200 mg by mouth once daily for 24 weeks.
Period: Overall Study
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Started | 50 | 49
Completed | 35 | 39
Not Completed | 15 | 10
Not completed — Lost to Follow-up | 1 | 3
Not completed — Off study Treatment | 9 | 3
Not completed — Poor scan quality | 3 | 2
Not completed — Missed Scan | 2 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate | Total
Number analyzed (Participants) | 35 | 39 | 74
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 35 | 39 | 74
  >=65 years | 0 | 0 | 0
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 46 [37 to 50] | 45 [38 to 51] | 45 [38 to 51]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 9 | 17
  Male | 27 | 30 | 57
Race/Ethnicity, Customized [Number; unit: participants]
  White, non-Hispanic | 15 | 15 | 30
  Black, non-Hispanic | 5 | 6 | 11
  Hispanic, regardless of race | 15 | 17 | 32
  American Indian, Alaskan Native | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 35 | 39 | 74
Current Smoker [Number; unit: participants]
  Yes | 10 | 16 | 26
  No | 25 | 23 | 48
10 year Coronary Heart Disease (CHD) risk [Median (Inter-Quartile Range); unit: 10yr Framingham CHD risk (%)] | 3 [1 to 6] | 3 [1 to 10] | 3 [1 to 8]
Relative FMD [Median (Inter-Quartile Range); unit: %] | 4.38 [2.88 to 6.76] | 3.93 [2.61 to 8.05] | 4.21 [2.76 to 6.76]
Baseline Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Niacin + Aspirin N=34; Fenofibrate N=39.
  mg/dL | 185 [171 to 212] | 184 [159 to 211] | 184 [165 to 211]
Triglycerides [Median (Inter-Quartile Range); unit: mg/dL] — Niacin + Aspirin N=34; Fenofibrate N=39.
  mg/dL | 254 [198 to 360] | 206 [171 to 293] | 232 [176 to 308]
High Density Lipoprotein (HDL)-Cholesterol [Number; unit: participants]
  Very low HDL-C (< 30 mg/dL (Men)/< 40 mg/dL (W)) | 10 | 12 | 22
  Low HDL-C (30-40 mg/dL (Men)/40-50 mg/dL (Women)) | 25 | 27 | 52
Men: HDL Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Since the eligibility requirements for HDL cholesterol differed for men and women, HDL cholesterol is reported separately for men and women.
  Niacin + Aspirin N=27; Fenofibrate N=30.
  mg/dL | 32 [30 to 35] | 36 [29 to 39] | 33 [30 to 37]
Women: HDL Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Since the eligibility requirements for HDL cholesterol differed for men and women, HDL cholesterol is reported separately for men and women.
  Niacin + Aspirin N=7; Fenofibrate N=9.
  mg/dL | 37 [36 to 49] | 38 [35 to 42] | 38 [36 to 46]
HDL Particles [Median (Inter-Quartile Range); unit: nmol/L] | 31.8 [28.4 to 35.4] | 30.2 [26.7 to 33.2] | 31.3 [27.2 to 34.8]
Non-HDL Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Niacin + Aspirin N=34; Fenofibrate N=39.
  mg/dL | 150 [135 to 169] | 153 [123 to 175] | 150 [128 to 169]
Low Density Lipoprotein (LDL) Cholesterol [Median (Inter-Quartile Range); unit: mg/dL] — Niacin + Aspirin N=29; Fenofibrate N=36.
  mg/dL | 103 [88 to 117] | 101 [84 to 120] | 103 [86 to 119]
Small LDL Particles [Median (Inter-Quartile Range); unit: nmol/L] | 1018 [803 to 1133] | 1052 [823 to 1222] | 1022 [816 to 1161]
Large HDL Particles [Median (Inter-Quartile Range); unit: nmol/L] | 2.1 [1.4 to 3.2] | 2.6 [1.5 to 3.7] | 2.5 [1.5 to 3.3]
HOMA-IR (Homeostatic model assessment - Insulin Resistance) [Median (Inter-Quartile Range); unit: HOMA IR Score] — Niacin + Aspirin N=34; Fenofibrate N=39.
  HOMA IR Score | 2.5 [1.9 to 4.5] | 3.2 [2.6 to 5.3] | 3.1 [2.1 to 4.8]
Interleukin(IL)-6 [Median (Inter-Quartile Range); unit: pg/ml] — Niacin + Aspirin N=34; Fenofibrate N=35.
  pg/ml | 1.1 [0.8 to 2.2] | 1.5 [0.8 to 2.2] | 1.3 [0.8 to 2.2]
C-reactive protein [Median (Inter-Quartile Range); unit: ug/ml] | 1.9 [1.0 to 5.4] | 1.5 [0.7 to 3.9] | 1.7 [0.8 to 4.3]
D-Dimer [Median (Inter-Quartile Range); unit: ug/ml] | 0.30 [0.22 to 0.37] | 0.25 [0.19 to 0.46] | 0.29 [0.19 to 0.42]

OUTCOME MEASURES:

1. Primary Outcome: Absolute Change in Relative FMD (%)
Description: The absolute change in maximum relative flow mediated dilation (FMD) (%) of the brachial artery from baseline to week 24.
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: % FMD
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 35 | 39
% FMD | 0.60 [-1.58 to 2.28] | 0.50 [-0.97 to 2.98]
Statistical Analysis 1: Comparison: Arm A: Extended-release Niacin With Aspirin; Test type: Superiority or Other; p = 0.28, Sign test; Stratified exact Wilcoxon signed rank test. Stratified by screening HDL-C level and statin use within 90 days prior to study entry
Statistical Analysis 2: Comparison: Arm B: Fenofibrate; Test type: Superiority or Other; p = 0.19, Sign test; [statistical method as in outcome 1, analysis 1]

2. Secondary Outcome: Change in Cholesterol
Description: Absolute change in total cholesterol from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan and had lipid panels at weeks 0 and 24.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 34 | 39
mg/dL | -9 [-26 to 3] | -2 [-28 to 25]

3. Secondary Outcome: Change in Triglycerides
Description: Change in Triglycerides (mg/dL) from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 34 | 39
mg/dL | -65 [-163 to 8] | -54 [-113 to -10]

4. Secondary Outcome: Men: Change in HDL Cholesterol
Description: Among men, change in HDL Cholesterol (mg/dL) from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: Men in the as-treated analysis population, limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 27 | 30
mg/dL | 3 [0 to 9] | 6.5 [0 to 12]

5. Secondary Outcome: Women: Change in HDL Cholesterol
Description: Among women, change in HDL cholesterol (mg/dL) from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: Women in the as-treated analysis population, limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 7 | 9
mg/dL | 16 [-1 to 22] | 8 [5 to 13]

6. Secondary Outcome: Change in HDL Particles
Description: Change in total HDL particles from week 0 to week 24
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 35 | 39
nmol/L | -1.7 [-4.3 to 2.1] | 4.3 [1.8 to 7.2]

7. Secondary Outcome: Change in Non-HDL Cholesterol
Description: Change in non-HDL Cholesterol (mg/dL) from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 34 | 39
mg/dL | -17 [-29 to 4] | -4 [-28 to 17]

8. Secondary Outcome: Change in LDL Cholesterol
Description: Change in LDL cholesterol (mg/dL) from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 27 | 35
mg/dL | -1 [-14 to 12] | 7 [-13 to 26]

9. Secondary Outcome: Change in Small LDL Particles
Description: Change in Small LDL particles from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 35 | 39
nmol/L | -176 [-410 to -19] | -119 [-320 to -17]

10. Secondary Outcome: Change in Large HDL Particles
Description: Change in Large HDL Particles from week 0 to week 24
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: nmol/L
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 35 | 39
nmol/L | 0.9 [0.1 to 3.3] | -0.3 [-0.9 to 0.5]

11. Secondary Outcome: Change in HOMA-IR
Description: Absolute change from week 0 to week 24 in insulin resistance as estimated by HOMA-IR
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: HOMA IR Score
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 34 | 35
HOMA IR Score | 1.3 [0.0 to 3.0] | 0.3 [-1.2 to 1.2]

12. Secondary Outcome: Change in IL-6
Description: Change in IL-6 from week 0 to week 24
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: pg/ml
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 32 | 33
pg/ml | 0.1 [-1.1 to 0.8] | 0.2 [-0.7 to 1.1]

13. Secondary Outcome: Change in C-reactive Protein (CRP)
Description: Change in C-reactive protein from week 0 to week 24.
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 35 | 39
ug/ml | -0.6 [-3.0 to 2.6] | 0.7 [-2.1 to 2.7]

14. Secondary Outcome: Change in D-Dimer
Description: Change in D-Dimer from week 0 to week 24
Time Frame: 0 and 24 weeks
Population: This is an as-treated analysis limited to 74 participants who had 24 weeks of follow up and a useable week 24 scan.
Measure: Median (Inter-Quartile Range); unit: ug/ml
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Number analyzed (Participants) | 35 | 39
ug/ml | 0.06 [-0.08 to 0.20] | 0.06 [-0.19 to 0.27]

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from randomization to the date the participant went off study.
Description: Grade≥2 nausea, vomiting diarrhea, ulcers, abnormal bleeding/bruising, and lab values. Other Grade≥3 signs/symptoms and all s/sx or labs that lead to a change in study treatment regardless of grade. Diagnoses per ACTG criteria for clinical events & diseases. See DAIDS Table for Grading the Severity of Adult and pediatric AEs, V1.0.
Arm/Group | Arm A: Extended-release Niacin With Aspirin | Arm B: Fenofibrate
Serious Adverse Events (participants affected / at risk) | 1/50 | 0/49
Other Adverse Events (participants affected / at risk) | 47/50 | 34/49
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Extended-release Niacin With Aspirin (N=50) | Arm B: Fenofibrate (N=49)
Pancreatitis (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Extended-release Niacin With Aspirin (N=50) | Arm B: Fenofibrate (N=49)
Abdominal pain (Gastrointestinal disorders) | 3 | 1
Diarrhoea (Gastrointestinal disorders) | 3 | 0
Nausea (Gastrointestinal disorders) | 7 | 2
Vomiting (Gastrointestinal disorders) | 4 | 1
Fatigue (General disorders) | 3 | 0
Alanine aminotransferase increased (Investigations) | 8 | 7
Aspartate aminotransferase increased (Investigations) | 10 | 4
Blood alkaline phosphatase increased (Investigations) | 7 | 0
Blood bilirubin increased (Investigations) | 17 | 8
Blood cholesterol increased (Investigations) | 11 | 12
Blood creatinine increased (Investigations) | 1 | 8
Blood glucose decreased (Investigations) | 1 | 5
Blood glucose increased (Investigations) | 13 | 6
Blood phosphorus decreased (Investigations) | 2 | 4
Blood triglycerides increased (Investigations) | 2 | 3
Blood uric acid increased (Investigations) | 9 | 1
Low density lipoprotein increased (Investigations) | 5 | 5
Myalgia (Musculoskeletal and connective tissue disorders) | 5 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 4 | 2
Paraesthesia (Nervous system disorders) | 3 | 0
Pruritus generalised (Skin and subcutaneous tissue disorders) | 3 | 0
Flushing (Vascular disorders) | 15 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No